CLINICAL TRIAL: NCT06643000
Title: A Single-center, Real-world Study Aimed At Evaluating the Efficacy and Safety of 240 Mg/d Furmonertinib Combined with Bevacizumab and Pemetrexed in the Treatment of Advanced NSCLC with EGFRm and Leptomeningeal Metastasis.
Brief Title: Evaluating High-dose Furmonertinib with Bevacizumab and Pemetrexed for EGFRm NSCLC with Leptomeningeal Metastasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qiming Wang, Deputy Director of Internal Medicine, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA2024-690
Record Dates: First submitted 2024-10-14; First posted 2024-10-15 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer; Leptomeningeal Metastasis; EGFR Gene Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis | interventions — aflutinib; Bevacizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Triple therapy (Experimental): furmonertinib combined with bevacizumab and pemetrexed
  Interventions: Drug: furmonertinib

INTERVENTIONS:
Drug: furmonertinib — furmonertinib (240 mg/d,po) combined with bevacizumab (15 mg/kg, every 3 weeks, ivgtt) and pemetrexed (50 mg) intrathecal chemotherapy / pemetrexed (500 mg/m²) intravenous chemotherapy, administered every 3 weeks.
  Other Names: bevacizumab; pemetrexed

SUMMARY:
The primary objective of this clinical study is to evaluate the efficacy of high-dose furmonertinib combined with bevacizumab and pemetrexed (triple therapy) in the treatment of non-small cell lung cancer (NSCLC) with leptomeningeal metastasis and epidermal growth factor receptor mutation (EGFRm) through overall survival (OS). The secondary objectives are to further assess the efficacy of the triple therapy in patients with EGFRm and leptomeningeal metastasis, including time to treatment failure (TTF), leptomeningeal objective response rate (ORR-LM), and clinical response rate.The study will also evaluate the impact of the triple therapy on quality of life using the EORTC QLQ-C30 scale and assess the safety of the therapy in EGFRm NSCLC patients with leptomeningeal metastasis, focusing primarily on adverse events and their severity (graded according to CTCAE v5.0), as well as their frequency.The exploratory objectives are to assess changes in intracranial pressure and the improvement rate of cerebrospinal fluid (CSF) before and after the triple therapy treatment. Additionally, the study will compare the genomic and epigenomic profile changes in circulating tumor DNA (ctDNA) from peripheral blood and cell-free DNA (cfDNA) from cerebrospinal fluid before and after treatment, and analyze their correlation with clinical outcomes, drug efficacy, and other clinical indicators.

The primary endpoint of this study is overall survival (OS). The secondary endpoints include time to treatment failure (TTF), leptomeningeal objective response rate (ORR-LM), clinical response rate, and quality of life assessment (EORTC QLQ-C30).The safety endpoints are adverse events and their severity (graded according to CTCAE v5.0), as well as the frequency of occurrence.

A total of 60 patients are planned to be enrolled, targeting eligible advanced NSCLC patients with EGFR mutations and leptomeningeal metastasis.

The intervention consists of furmonertinib (240 mg/d, po) combined with bevacizumab (15 mg/kg, every 3 weeks, ivgtt) and pemetrexed (50 mg) intrathecal chemotherapy / pemetrexed (500 mg/m²) intravenous chemotherapy, administered every 3 weeks.

DETAILED DESCRIPTION:
Leptomeningeal metastasis (LM) is a fatal complication of advanced lung cancer. In recent years, with the rapid advancement of precision therapy for lung cancer, the survival time of patients with advanced lung cancer has significantly increased, leading to a rapid rise in the incidence of LM. It is reported that the incidence of LM in patients with advanced non-small cell lung cancer (NSCLC) reaches 3%-5%, and as high as 9.4% among patients with epidermal growth factor receptor (EGFR) mutations. The prognosis of NSCLC patients with LM is extremely poor, with a median overall survival (OS) of only 4-6 weeks without treatment[1]. Due to the presence of the blood-brain barrier (BBB), which limits drug penetration, as well as the efflux mechanisms of transport proteins on the BBB, effectively treating patients with LM remains a significant challenge.

For brain or leptomeningeal metastases driven by genetic mutations, both the Lung Cancer Brain (Leptomeningeal) Metastasis Diagnosis and Treatment Consensus (2017) and the 2024 NCCN Guidelines recommend tyrosine kinase inhibitors (TKIs) as the first-line treatment. Most studies on first- and second-generation EGFR-TKIs for leptomeningeal metastasis are retrospective and show relatively limited efficacy. Pulse dosing of erlotinib appears to achieve relatively longer overall survival (OS), but both studies included only a few patients. In two prospective studies on afatinib and gefitinib, OS did not exceed four months. The BLOOM study included 41 patients with CSF-confirmed EGFR-mutant NSCLC with leptomeningeal metastasis who received osimertinib at a dose of 160 mg/d. The LM objective response rate (ORR) was 62%, progression-free survival (PFS) was 8.6 months, and OS was 11.0 months. While the overall efficacy showed room for improvement, safety concerns were notable: 66% of patients experienced grade 3 or higher adverse events, 51% experienced serious adverse events (SAEs), 22% discontinued treatment due to adverse events, and 12% required dose reduction. In summary, improving clinical outcomes for patients with EGFR-mutant NSCLC with LM, while reducing toxicity, remains a key area for further exploration.

Furmonertinib (brand name: Aifisha, formerly known as alflutinib/AST2818) is a third-generation EGFR TKI independently developed by Shanghai Allist Pharmaceuticals. Furmonertinib has demonstrated strong antitumor activity and manageable safety characteristics in advanced patients with EGFR exon 20 T790M point mutations (T790M-positive). It was approved by the NMPA in March 2020. In June 2022, furmonertinib received approval from the National Medical Products Administration (NMPA) for first-line treatment of adult patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring EGFR exon 19 deletions or exon 21 (L858R) substitution mutations.

In the Phase I-IIa study, furmonertinib demonstrated good tolerability, with no dose-related toxic reactions observed across the dose groups ranging from 20 mg to 240 mg. At a dose of 240 mg/day, the safety and tolerability were favorable, with an incidence of ≥ Grade 3 adverse events (AEs) at 11%, and serious adverse events occurring in 11% of patients. Dose reduction due to AEs occurred in 6% of patients, and no patients discontinued treatment due to AEs. The most common adverse reactions included diarrhea (33%), rash (33%), decreased white blood cell count (28%), elevated serum creatinine (22%), and proteinuria (22%), all of which were Grade 1-2. The most frequent ≥ Grade 3 AE was elevated ALT (6%). Overall, the drug was well-tolerated, and adverse events were relatively manageable.

An Ib phase clinical study named FAVOUR enrolled 30 patients with advanced NSCLC harboring EGFR Exon20ins mutations, who received furmonertinib at doses of 160 mg/day or 240 mg/day. Data from the initial treatment cohort of 10 patients receiving 240 mg/day of furmonertinib have been released. The results showed that the objective response rate (ORR) assessed by independent review committee (IRC) reached 60%, the disease control rate (DCR) was 100%, and progression-free survival (PFS) has not yet been reached. Additionally, safety was favorable, with no reports of ≥ Grade 3 adverse events, suggesting that high-dose furmonertinib holds promise for the treatment of patients with EGFR uncommon mutations.

In addition to showing good efficacy in patients with advanced NSCLC harboring classic and uncommon EGFR mutations, furmonertinib has also demonstrated promising central nervous system (CNS) activity. Preclinical studies indicated that 24 hours after administration in animal models, the ratio of furmonertinib's prototype drug and its major active metabolite AST2818 in brain tissue AUC0-24h to plasma AUC0-24h was greater than 1, suggesting that furmonertinib can penetrate the blood-brain barrier (BBB). In its Phase IIb clinical study, furmonertinib achieved a CNS objective response rate (ORR) of 66%, CNS disease control rate (DCR) of 100%, and CNS progression-free survival (PFS) of 11.6 months in patients with EGFR T790M mutation and brain metastases. Additionally, in its Phase I/II study, CNS efficacy increased with higher doses: the 80 mg/day dose achieved a CNS ORR of 60% and a CNS PFS of 9.7 months, while the 160 mg/day dose resulted in a CNS ORR of 84.6% and a CNS PFS of 19.3 months . For patients with refractory leptomeningeal metastasis (LM), increasing the dose of furmonertinib may offer enhanced antitumor activity.

Based on the above findings, researchers conducted a real-world study, and data analysis revealed that furmonertinib at a dose of 240 mg/day demonstrated significant efficacy in the treatment of leptomeningeal metastasis, with patients overall showing good tolerability. From May 2021 to December 2023, a total of 48 patients were enrolled, of which 35 patients had an ECOG performance status ≥3, accounting for 72.9%. Of these, 35 patients (72.9%) had previously received other third-generation EGFR-TKI treatments. Seventeen patients (35.4%) were treated with furmonertinib monotherapy. The median follow-up time was 15 months. The median overall survival (OS) was 8.433 months (95% CI, 5.481-11.386 months), and the median time to treatment discontinuation (TTD) was 8.267 months (95% CI, 5.395-11.138 months). The clinical response rate was 75%. According to the RANO-LM radiological criteria, the leptomeningeal metastasis (LM) objective response rate (ORR) and disease control rate (DCR) were 50.0% and 92.1%, respectively. The treatment was well tolerated overall, consistent with previous reports. Twenty-two patients (45.8%) experienced treatment-related adverse events (TRAEs), and three patients (6.3%) experienced ≥ Grade 3 TRAEs. The investigators found that high-dose TKI monotherapy improved prognosis in patients with leptomeningeal metastasis, but the median OS still did not exceed one year. Further exploration is needed to extend survival in these patients, and more treatment modalities are currently under investigation.

In terms of systemic combination therapy, studies have shown that bevacizumab can enhance the penetration of TKIs into cerebrospinal fluid, increasing their concentration in brain tissue. A retrospective analysis of 27 patients receiving osimertinib combined with bevacizumab showed that the median OS in the combination group (n=16) and the monotherapy group (n=11) was 18.0 months and 13.7 months (p = 0.046), respectively, and intracranial PFS (iPFS) was 10.6 months and 5.5 months (p = 0.037) . These results suggest that osimertinib combined with bevacizumab may significantly improve the median OS and intracranial PFS in patients with leptomeningeal metastasis compared to osimertinib monotherapy. Additionally, combining intrathecal chemotherapy to increase local drug concentration can improve efficacy and survival benefits. An I/II phase study showed that intrathecal injection of pemetrexed achieved good efficacy in lung cancer patients with leptomeningeal metastasis who had failed multiple lines of targeted therapy: the ORR was 84.6%, and the median OS was 9 months. Among patients who achieved a clinical response (CR or PR), the median OS was 12 months, and the safety profile was significantly better than with traditional drugs . When pemetrexed was administered intravenously in combination with systemic therapy, patients also benefited in terms of survival. A retrospective study of 110 patients with EGFR-mutant advanced NSCLC treated with EGFR TKIs found that after leptomeningeal metastasis, patients who received systemic pemetrexed chemotherapy had a longer overall survival than those who did not (13.7 vs 4.0 months, p = 0.008) .

Based on the above findings, this study aims to explore the efficacy and safety of furmonertinib 240 mg/day combined with bevacizumab and pemetrexed in EGFR-mutant NSCLC patients with leptomeningeal metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Have obtained written informed consent from the patient or his or her legal representative;
2. The patient is ≥18 years old, male or female;
3. Non-small cell lung cancer confirmed by histological or cytological pathology;
4. Genetic testing confirming positive for classical or non-classical EGFR mutations;
5. After comprehensive clinical evaluation according to the "EANO-ESMO" meningeal metastasis diagnostic criteria, the comprehensive clinical evaluation of patients with definite meningeal metastasis included symptom evaluation, imaging evaluation, and/or cerebrospinal fluid pathology evaluation;
6. Patients with newly diagnosed leptomeningeal metastases and those with disease progression after previous antineoplastic therapy were eligible;
7. ECOG Performance Status 0-3;
8. Prior treatment with radiation or surgery targeting the central nervous system is permitted;
9. Admit patients with CNS symptoms or signs, but those symptoms or signs are not life threatening;
10. Fertile men or women with the possibility of becoming pregnant must use a highly effective method of contraception (such as oral contraceptives, intrauterine devices, abstinence or barrier contraception combined with spermicides) during the course of the trial and continue contraception for 12 months after the end of treatment.

Exclusion Criteria:

* 1)Patients currently have tumors other than NSCLC; 2)Have had or have a history of other malignancies within the last 5 years, other than basal cell carcinoma of the skin, carcinoma in situ of the cervix, and ductal carcinoma in situ of the breast that have been effectively controlled; 3)Serious digestive tract diseases that affect drug use and absorption, including but not limited to peptic ulcer, inflammatory bowel disease, etc.

  4)Evidence of any severe or uncontrolled systemic disease, including uncontrolled hypertension, diabetes, and active bleeding, any that the investigator deems to be detrimental to the patient's participation in the study or to adherence to the protocol, or active infections including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV); 5)A history of interstitial lung disease, drug-induced interstitial lung disease, prior history of radiation pneumonia requiring steroid treatment, or any evidence of active interstitial lung disease; 6)The presence of significant arrhythmias (such as prolonged QT interval > 500ms) or heart failure (left ventricular ejection fraction < 50%) 7)Pregnant or lactating women; 8)Patients who received a live vaccine within 4 weeks before treatment began; 9)Patients who are or have been involved in another clinical study within 4 weeks; 10)Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that, in the investigator's opinion, may increase the risks associated with participating in the study or may interfere with the interpretation of the study results; Or subjects who may not be able to complete the study or comply with the requirements of the study (for administrative or other reasons).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
OS | the time between the date of enrollment and the date of death from any cause
  overall survive time

SECONDARY OUTCOMES:
TTF | The time interval from the start of the triple therapy to treatment failure
  time to treatment failure
ORR-LM | the proportion of patients whose leptomeningeal lesions achieve a complete response (CR) or partial response (PR) during the study period from the first administration of the study drug until leptomeningeal disease progression
  Objective Response Rate in Leptomeningeal Metastases
CRR | the proportion of patients whose CR, OR, or PR lasts for at least one week
  Clinical response rate

CONTACTS AND LOCATIONS:
Overall Officials: Qiming Wang, MD, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No